CLINICAL TRIAL: NCT06214767
Title: Study on Treatment Decision-Making and Prognostic Follow-Up for Untreated Cerebral Cavernous Malformations
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: RenJi Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other); Guangzhou Red Cross Hospital (Other); Affiliated Hospital of Guangdong Medical University (Other); Shanxi Provincipal People's Hospital (Unknown); Qilu Hospital of Shandong University (Other); Second Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: HX-B-2023058
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hemangioma, Cavernous, Central Nervous System
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate and predict the risk associated with cerebral cavernous malformations (CCMs) using advanced artificial intelligence and radiomics analysis technology. The study focuses on individuals who have been diagnosed with cerebral cavernous malformations (CCMs).

Main Questions to Answer:

How can AI-based radiomics features predict the risk of complications (such as bleeding or epilepsy) in individuals with CCMs? What are the most reliable imaging and clinical markers for assessing the prognosis of CCMs? Participants will be required to undergo regular medical imaging to gather traditional and radiomics imaging features.

Participants will provide clinical data, including past medical history and results of any laboratory tests.

Participants will be part of a three-year follow-up observation to monitor the progression or stability of CCMs.

Contribution of biological samples for advanced testing might also be requested.

This study aims to create an AI-based decision-making tool that will guide clinicians in the management of CCM, with the potential to significantly improve patient outcomes through personalized medical approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CCM based on brain MRI (T1, T2, SWI, and T2-Fluid-Attenuated Inversion Recovery).
2. Patients who have not received invasive treatment (surgery, radiotherapy, or multimodal therapy) in the past.
3. Patients undergoing surgery, or their legal guardians, agree to collect lesion tissue samples for related studies and sign a consent form for the collection of biological samples.
4. Patients under conservative observation, or their legal guardians, agree to collect imaging data for related research and sign a consent form for the use of imaging data.
5. Willingness to participate in long-term follow-up.

Exclusion Criteria:

1. Patients with acute intracranial symptomatic hemorrhage requiring emergency surgery.
2. Patients with other intracranial diseases, such as aneurysms, tumors, or other vascular malformations, excluding developmental venous anomalies (DVA).
3. Patients with severe underlying diseases affecting their functional status and short-term life expectancy.
4. Patients with severe psychiatric or psychological disorders.
5. Incomplete clinical or imaging data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Untreated cerebral cavernous malformation patients
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome:mRS | 3 years
  Last follow-up with a modified Rankin Scale (mRS) score greater than 2 persisting for at least one year

SECONDARY OUTCOMES:
Radiological Outcome:Bleeding | 3 years
  Bleeding is defined as the presence of new hemorrhage identified on radiological imaging in patients.
Radiological Outcome:Increase in lesion volume | 3 years
  An increase in lesion volume is defined as a 20% or more increase in the size of the lesion, as shown by follow-up imaging compared to previous measurements.
Syndrome Outcome:Drug-resistant epilepsy | 3 years
  Epilepsy is considered drug-resistant when a person has failed to achieve sustained seizure freedom despite adequate trials of two appropriate and well-tolerated antiepileptic drug regimens, either as monotherapies or in combination.
Syndrome Outcome:Focal neurological deficits | 3 years
  Focal neurological deficits can manifest as weakness, numbness, loss of coordination, or changes in sensation specific to the affected area, and are typically indicative of underlying neurological conditions or injuries.
All-cause mortality | 3 years
  All-cause mortality refers to the proportion of deaths due to any cause within the follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided